CLINICAL TRIAL: NCT01408888
Title: Study to Evaluate the Effect of LY2189265 on Sitagliptin Pharmacokinetics in Patients With Type 2 Diabetes Mellitus
Brief Title: A Study of LY2189265 and Sitagliptin in Participants With Type 2 Diabetes
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 14361; H9X-MC-GBDW (Other: Eli Lilly and Company)
Record Dates: First submitted 2011-08-02; First posted 2011-08-03 (Estimated); Results first posted 2014-10-07 (Estimated); Last update posted 2014-10-07 (Estimated); Status verified 2014-10

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — dulaglutide; Sitagliptin Phosphate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- LY2189265, Sitagliptin + LY2189265 (Experimental): A single 1.5-milligram (mg) dose of LY2189265 administered subcutaneously (Treatment 1). There was a washout period of at least 21 days before crossing over and receiving 100 mg of sitagliptin administered orally, once daily for 18 days in combination with two separate single 1.5-mg doses of LY2189265 administered subcutaneously, immediately prior to the sitagliptin doses on Day 5 and Day 12 (Treatment 2).
  Interventions: Biological: LY2189265; Drug: Sitagliptin
- Sitagliptin + LY2189265, LY2189265 (Experimental): 100 mg of sitagliptin administered orally, once daily for 18 days in combination with two separate single 1.5-mg doses of LY2189265 administered subcutaneously, immediately prior to the sitagliptin doses on Day 5 and Day 12 (Treatment 2). There was a washout of at least 21 days before crossing over and receiving a single 1.5 mg dose of LY2189265 administered subcutaneously (Treatment 1).
  Interventions: Biological: LY2189265; Drug: Sitagliptin

INTERVENTIONS:
Biological: LY2189265 — Administered subcutaneously
  Other Names: Dulaglutide
Drug: Sitagliptin — Administered orally

SUMMARY:
The purpose of this study is to study the effect of LY2189265 on how the body absorbs and processes a Type 2 Diabetes Mellitus (T2DM) drug (sitagliptin) and how sitagliptin affects LY2189265 when they are taken together.

The duration of participation in this study is expected to be approximately 61 days. The study requires 2 clinic confinements (one of 2 nights and one of 19 nights duration).

The study involves 3 injections, subcutaneous, of 1.5 milligrams (mg) LY2189265 and 18 daily doses of 100 mg sitagliptin tablets administered orally.

ELIGIBILITY:
Inclusion Criteria:

* are males or females, diagnosed with T2DM (Type 2 Diabetes Mellitus) for ≥3 months prior to screening
* male participants with female partners of child-bearing potential, or partners who are pregnant or breastfeeding, agree to use a reliable method of contraception from the time of the first dose until 3 months after the last dose of investigational product, as determined by the investigator. The method may be one of the following:

  * condom with spermicidal agent
  * male participant sterilization
  * true abstinence (which is in line with the participant's usual lifestyle choice; withdrawal or calendar methods are not considered acceptable)
* female participants not of child-bearing potential (that is, are postmenopausal or permanently sterilized [such as, tubal occlusion, hysterectomy, bilateral salpingectomy]). Such participants will not be required to use contraception but must test negative for pregnancy at the time of enrollment. Postmenopausal is defined as at least 1 year post cessation of menses (without an alternative medical cause) or at least 1 year of spontaneous amenorrhea, with follicle stimulating hormone (FSH) ≥40 milli-international units/milliliter (mIU/mL)
* female participants who have undergone sterilization by tubal ligation: agree to use a condom in conjunction with spermicidal gel, foam, cream, film or suppository from the time of screening until 3 months after the last dose of investigational product. Such participants must also test negative for pregnancy at the time of enrollment
* have a body mass index (BMI) of between 23.0 and 40.0 kilograms/meter squared (kg/m^2), inclusive, at the time of screening
* have T2DM controlled with diet and exercise alone, or are on a stable dose of metformin Immediate Release (IR) for at least 4 weeks prior to screening, or are on metformin Extended Release (ER) and are capable/willing to be switched onto metformin IR or washed out prior to the first dose of investigational product, or are on sulfonylureas, acarbose (or other disaccharidase inhibitors), thiazolidinediones, or meglitinides and are capable/willing to be washed out prior to the first dose of investigational product
* have a fasting blood glucose value at screening ≤15.3 millimoles/liter (mmol/L) (275 milligrams/deciliter [mg/dL])
* have a glycosylated hemoglobin A1c (HbA1c) value at screening (or within 4 weeks prior to screening) of 6.5% to 10%
* have clinical laboratory test results within normal reference range for the population or within normal reference range for the investigator site, or results with acceptable deviations that are judged to be not clinically significant by the investigator. Abnormalities of serum glucose, serum lipids, urinary glucose, and urinary protein consistent with T2DM are acceptable.
* have creatinine clearance (CrCl) of greater than 50 milliliters/minute (mL/min) at screening estimated by the Cockcroft-Gault formula
* have venous access sufficient to allow for blood sampling as per the protocol
* are reliable and willing to make themselves available for the duration of the study and are willing to follow study procedures

Exclusion Criteria:

* are currently enrolled in, have completed or discontinued within the last 30 days from, a clinical trial involving an investigational product, or are concurrently enrolled in any other type of medical research judged not to be scientifically or medically compatible with this study
* have known allergies to glucagon-like-peptide 1 (GLP-1)-related compounds, including LY2189265 or to sitagliptin-related compounds or any components of either formulation
* are persons who have previously completed or withdrawn from this study or any other study investigating LY2189265 in the 3 months prior to screening or have received glucagon-like peptides or incretin mimetics in the 3 months prior to screening
* have taken insulin, chlorpropamide, or alpha-glucosidase inhibitors within 30 days prior to screening
* have an abnormality in the 12-lead electrocardiogram (ECG) that, in the opinion of the investigator, increases the risks associated with participating in the study
* have poorly controlled hypertension (systolic blood pressure [BP] >160 millimeters of mercury [mmHg] and/or diastolic BP >100 mmHg) and/or evidence of labile BP including symptomatic postural hypotension
* have a history or presence of respiratory, hepatic, renal, endocrine, hematological, or neurological disorders capable of significantly altering the absorption, metabolism, or elimination of drugs; of constituting a risk when taking the study medication; or of interfering with the interpretation of data
* have a history or presence of cardiovascular disorder (including myocardial infarction, cerebrovascular accident, venous thromboembolism, arrhythmia [judged by the investigator to be clinically significant], or angina) within the last year, have symptoms or signs of congestive heart failure, or are expected to require coronary artery bypass surgery or angioplasty
* have a history or presence of pancreatitis (history of chronic pancreatitis or idiopathic acute pancreatitis) or gastrointestinal disorder, for example relevant esophageal reflux or gall bladder disease, or any gastrointestinal disease which impacts gastric emptying (GE) (such as, gastric bypass surgery, pyloric stenosis, with the exception of appendectomy) or could be aggravated by GLP-1 analogs or dipeptidyl peptidase-4 (DPP-4) inhibitors. Participants with dyslipidemia, and participants who had cholecystolithiasis (removal of gall stones) and/or cholecystectomy (removal of gall bladder) in the past, with no further sequelae, may be included in the study at the discretion of the screening physician
* have any existing medical condition that might interfere with interpretation of the data, including a history of gastrointestinal surgery (with the exception of appendectomy performed more than 12 months ago), peptic ulceration, gastrointestinal bleeding, diabetic gastroparesis, ulcerative colitis, Crohn's disease, Irritable Bowel Syndrome (IBS), gastric bypass, or laparoscopic gastric banding
* show evidence of significant active neuropsychiatric disease
* have had 2 or more episodes of severe hypoglycemia within the last 6 months prior to screening
* have personal or family history of medullary thyroid cancer (MTC) or a genetic condition that predisposes to MTC
* regularly uses known drugs of abuse and/or show positive findings on urinary drug screening
* intend to start new concomitant medication during the study, including over-the-counter and herbal medication, regularly use drugs that directly reduce gastrointestinal motility and/or regularly use systemic corticosteroids by oral, intravenous, or intramuscular route, or potent, inhaled, or intranasal steroids known to have a high rate of systemic absorption
* show evidence of human immunodeficiency virus (HIV) infection and/or positive human HIV antibodies
* show evidence of hepatitis C and/or positive hepatitis C antibody
* show evidence of hepatitis B and/or positive hepatitis B surface antigen
* have donated blood of more than 500 milliliters (mL) within the last month prior to screening
* have an average weekly alcohol intake that exceeds 21 units per week (males up to age 65) and 14 units per week (males over 65 and females), or are unwilling to stop alcohol consumption from Day -3 of each period until after the last pharmacokinetic (PK) sample has been taken for that period, or to limit alcohol intake to a maximum of 2 units/day on all other days from screening through to follow-up. (1 unit = 12 ounces [oz] or 360 mL of beer; 5 oz or 150 mL of wine; 1.5 oz or 45 mL of distilled spirits)
* smoke more than 10 cigarettes (or equivalent in nicotine) per day, and are unwilling to refrain from smoking on the day of LY2189265/sitagliptin administration or are unable to abide by Clinical Research Unit (CRU) restrictions on other inpatient days
* are participants who, in the opinion of the investigator, are in any way unsuitable to participate in the study
* have any medical conditions, medical history or are taking any medication which are contraindicated

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2011-08; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (3):
- United States (3):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Daytona Beach, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Honolulu, Hawaii
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Dallas, Texas

RESULTS

PARTICIPANT FLOW:
Groups:
- LY2189265, Sitagliptin + LY2189265: First Intervention Period: A single 1.5-milligram (mg) subcutaneous (SC) injection of LY2189265 on Day 1 (Treatment 1).
  Second Intervention Period: 100 mg of sitagliptin, administered orally, once daily on Day 1 to Day 18 with single SC injections of 1.5 mg LY2189265 immediately prior to the sitagliptin dose on Day 5 and Day 12 (Treatment 2).
  There was a washout of at least 21 days between treatments.
- Sitagliptin + LY2189265, LY2189265: First Intervention Period: 100 mg of sitagliptin, administered orally, once daily on Day 1 to Day 18 with single SC injections of 1.5 mg LY2189265 immediately prior to the sitagliptin dose on Day 5 and Day 12 (Treatment 2).
  Second Intervention Period: A single 1.5-mg SC injection of LY2189265 on Day 1 (Treatment 1).
  There was a washout of at least 21 days between treatments.
Period: First Intervention
Arm/Group | LY2189265, Sitagliptin + LY2189265 | Sitagliptin + LY2189265, LY2189265
Started | 18 | 11
Received at Least 1 Dose of Drug | 18 | 11
Completed | 18 | 8
Not Completed | 0 | 3
Not completed — Adverse Event | 0 | 1
Not completed — Withdrawal by Subject | 0 | 2
Period: Washout of at Least 21 Days
Arm/Group | LY2189265, Sitagliptin + LY2189265 | Sitagliptin + LY2189265, LY2189265
Started | 18 | 8
Completed | 18 | 8
Not Completed | 0 | 0
Period: Second Intervention
Arm/Group | LY2189265, Sitagliptin + LY2189265 | Sitagliptin + LY2189265, LY2189265
Started | 18 | 8
Completed | 16 | 8
Not Completed | 2 | 0
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Adverse Event | 1 | 0

BASELINE CHARACTERISTICS:
Population: Participants who received at least one dose of study drug (LY2189265 or Sitagliptin).
Groups:
- Entire Study Population: Participants who received at least one dose of study drug (LY2189265 or Sitagliptin).
Arm/Group | Entire Study Population
Number analyzed (Participants) | 29
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.7 (11.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 19
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5
  Not Hispanic or Latino | 24
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 4
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 14
  White | 11
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 29

OUTCOME MEASURES:

1. Primary Outcome: Pharmacokinetics: Area Under the Concentration Versus Time Curve (AUC) of Sitagliptin
Description: Area under the sitagliptin pharmacokinetic (PK) concentration versus time curve (AUC [0-tau]) during one dosing interval (24 hours) is summarized.
Time Frame: Predose and up to 24 hours postdose on Day 4, Day 6, and Day 13 of Treatment 2
Population: Participants who received at least one dose of sitagliptin with evaluable sitagliptin AUC data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms times hour/milliliter(ng*h/mL)
Groups:
- 100 mg Sitagliptin (Day 4): Sitagliptin + LY2189265: 100 milligrams (mg) of sitagliptin, administered orally, once daily on Day 1 to Day 18 with single subcutaneous (SC) injections of 1.5 mg LY2189265 immediately prior to the sitagliptin dose on Day 5 and Day 12 (Treatment 2). Measure taken at Day 4.
- 100 mg Sitagliptin + 1.5 mg LY2189265 (Day 6): Sitagliptin + LY2189265: 100 mg of sitagliptin, administered orally, once daily on Day 1 to Day 18 with single SC injections of 1.5 mg LY2189265 immediately prior to the sitagliptin dose on Day 5 and Day 12 (Treatment 2). Measure taken at Day 6.
- 100 mg Sitagliptin + 1.5 mg LY2189265 (Day 13): Sitagliptin + LY2189265: 100 mg of sitagliptin, administered orally, once daily on Day 1 to Day 18 with single SC injections of 1.5 mg LY2189265 immediately prior to the sitagliptin dose on Day 5 and Day 12 (Treatment 2). Measure taken at Day 13.
Arm/Group | 100 mg Sitagliptin (Day 4) | 100 mg Sitagliptin + 1.5 mg LY2189265 (Day 6) | 100 mg Sitagliptin + 1.5 mg LY2189265 (Day 13)
Number analyzed (Participants) | 28 | 29 | 26
nanograms times hour/milliliter(ng*h/mL) | 3210 (34) | 3240 (36) | 2970 (54)

2. Primary Outcome: Pharmacokinetics: Maximum Observed Drug Concentration (Cmax) of Sitagliptin
Time Frame: Predose and up to 24 hours postdose on Day 4, Day 6, and Day 13 of Treatment 2
Population: Participants who received at least one dose of sitagliptin with evaluable sitagliptin Cmax data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms/milliliter (ng/mL)
Groups:
- 100 mg Sitagliptin + 1.5 mg LY2189265 (Day 6): Sitagliptin + LY2189265: 100 mg of sitagliptin, administered orally, once daily on Day 1 to Day 18 with single SC injections of 1.5 mg of LY2189265 immediately prior to the sitagliptin dose on Day 5 and Day 12 (Treatment 2). Measure taken at Day 6.
Arm/Group | 100 mg Sitagliptin (Day 4) | 100 mg Sitagliptin + 1.5 mg LY2189265 (Day 6) | 100 mg Sitagliptin + 1.5 mg LY2189265 (Day 13)
Number analyzed (Participants) | 28 | 29 | 27
nanograms/milliliter (ng/mL) | 417 (46) | 374 (61) | 318 (77)

3. Secondary Outcome: Pharmacokinetics: Time of Maximum Observed Drug Concentration (Tmax) of Sitagliptin
Time Frame: Predose and up to 24 hours post dose on Day 4, Day 6, and Day 13 of Treatment 2
Population: Participants who received at least one dose of sitagliptin with evaluable sitagliptin tmax data
Measure: Median (Full Range); unit: hours
Arm/Group | 100 mg Sitagliptin (Day 4) | 100 mg Sitagliptin + 1.5 mg LY2189265 (Day 6) | 100 mg Sitagliptin + 1.5 mg LY2189265 (Day 13)
Number analyzed (Participants) | 28 | 29 | 27
hours | 1.00 [0.500 to 4.00] | 2.00 [0.500 to 16.0] | 2.00 [0.500 to 12.0]

4. Secondary Outcome: Pharmacokinetics: Area Under the Concentration Versus Time Curve (AUC) of LY2189265
Description: Area under the LY2189265 pharmacokinetic (PK) concentration versus time curve (AUC [0-tau]) during one dosing interval (168 hours) is summarized.
Time Frame: Predose and up to 168 hours postdose on Day 1 of Treatment 1 and on Day 5 and Day 12 of Treatment 2
Population: Participants who received at least one dose of LY2189265 with evaluable LY2189265 AUC data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms times hour/milliliter(ng*h/mL)
Groups:
- 1.5 mg LY2189265 (Day 1): Sitagliptin + LY2189265: A single, 1.5-milligram (mg) dose of LY2189265 administered subcutaneously (Treatment 1). There was a washout period of at least 21 days before crossing over and receiving 100 mg of sitagliptin administered orally, once daily for 18 days in combination with two separate single 1.5-mg doses of LY2189265 administered subcutaneously, immediately prior to the sitagliptin doses on Day 5 and Day 12 (Treatment 2). Measure taken on Day 1 of Treatment 1.
- 100 mg Sitagliptin + 1.5 mg LY2189265 (Day 5): Sitagliptin + LY2189265: A single, 1.5-mg dose of LY2189265 administered subcutaneously (Treatment 1). There was a washout period of at least 21 days before crossing over and receiving 100 mg of sitagliptin administered orally, once daily for 18 days in combination with two separate single 1.5-mg doses of LY2189265 administered subcutaneously, immediately prior to the sitagliptin doses on Day 5 and Day 12 (Treatment 2). Measure taken on Day 5 of Treatment 2.
- 100 mg Sitagliptin + 1.5 mg LY2189265 (Day 12): Sitagliptin + LY2189265: A single, 1.5-mg dose of LY2189265 administered subcutaneously (Treatment 1). There was a washout period of at least 21 days before crossing over and receiving 100 mg of sitagliptin administered orally, once daily for 18 days in combination with two separate single 1.5-mg doses of LY2189265 administered subcutaneously, immediately prior to the sitagliptin doses on Day 5 and Day 12 (Treatment 2). Measure taken on Day 12 of Treatment 2.
Arm/Group | 1.5 mg LY2189265 (Day 1) | 100 mg Sitagliptin + 1.5 mg LY2189265 (Day 5) | 100 mg Sitagliptin + 1.5 mg LY2189265 (Day 12)
Number analyzed (Participants) | 26 | 27 | 26
nanograms times hour/milliliter(ng*h/mL) | 6590 (40) | 8890 (26) | 13900 (26)

5. Secondary Outcome: Pharmacokinetics: Maximum Observed Drug Concentration (Cmax) of LY2189265
Time Frame: Predose and up to 168 hours postdose on Day 1 of Treatment 1 and on Day 5 and Day 12 of Treatment 2
Population: Participants who received at least one dose of LY2189265 with evaluable LY2189265 Cmax data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms/milliliter (ng/mL)
Groups:
- 1.5 mg LY2189265 (Day 1): Sitagliptin + LY2189265: A single, 1.5-mg dose of LY2189265 administered subcutaneously (Treatment 1). There was a washout period of at least 21 days before crossing over and receiving 100 mg of sitagliptin administered orally, once daily for 18 days in combination with two separate single 1.5 mg doses of LY2189265 administered subcutaneously, immediately prior to the sitagliptin doses on Day 5 and Day 12 (Treatment 2). Measure taken on Day 1 of Treatment 1.
- 100 mg Sitagliptin + 1.5 mg LY2189265 (Day 5): Sitagliptin + LY2189265: A single, 1.5-mg dose of LY2189265 administered subcutaneously (Treatment 1). There was a washout period of at least 21 days before crossing over and receiving 100 mg of sitagliptin administered orally, once daily for 18 days in combination with two separate single 1.5 mg doses of LY2189265 administered subcutaneously, immediately prior to the sitagliptin doses on Day 5 and Day 12 (Treatment 2). Measure taken on Day 5 of Treatment 2.
- 100 mg Sitagliptin + 1.5 mg LY2189265 (Day 12): Sitagliptin + LY2189265: A single, 1.5-mg dose of LY2189265 administered subcutaneously (Treatment 1). There was a washout period of at least 21 days before crossing over and receiving 100 mg of sitagliptin administered orally, once daily for 18 days in combination with two separate single 1.5 mg doses of LY2189265 administered subcutaneously, immediately prior to the sitagliptin doses on Day 5 and Day 12 (Treatment 2). Measure taken on Day 12 of Treatment 2.
Arm/Group | 1.5 mg LY2189265 (Day 1) | 100 mg Sitagliptin + 1.5 mg LY2189265 (Day 5) | 100 mg Sitagliptin + 1.5 mg LY2189265 (Day 12)
Number analyzed (Participants) | 26 | 29 | 26
nanograms/milliliter (ng/mL) | 52.9 (37) | 68.1 (25) | 101 (28)

6. Secondary Outcome: Pharmacokinetics: Time of Maximum Observed Drug Concentration (Tmax) of LY2189265
Time Frame: Predose and up to 168 hours postdose on Day 1 of Treatment 1 and on Day 5 and Day 12 of Treatment 2
Population: Participants who received at least one dose of LY2189265 with evaluable LY2189265 tmax data.
Measure: Median (Full Range); unit: hours
Groups:
- 1.5 mg LY2189265 (Day 1): Sitagliptin + LY2189265: A single, 1.5-mg dose of LY2189265 administered subcutaneously (Treatment 1). There was a washout period of at least 21 days before crossing over and receiving 100 mg of sitagliptin administered orally, once daily for 18 days in combination with two separate single 1.5-mg doses of LY2189265 administered subcutaneously, immediately prior to the sitagliptin doses on Day 5 and Day 12 (Treatment 2). Measure taken on Day 1 of Treatment 1.
Arm/Group | 1.5 mg LY2189265 (Day 1) | 100 mg Sitagliptin + 1.5 mg LY2189265 (Day 5) | 100 mg Sitagliptin + 1.5 mg LY2189265 (Day 12)
Number analyzed (Participants) | 26 | 29 | 26
hours | 72.0 [12.0 to 120] | 72.0 [48.0 to 144] | 59.8 [12.0 to 120]

ADVERSE EVENTS:
Groups:
- LY2189265: LY2189265: a single, 1.5-milligram (mg) dose of LY2189265 administered subcutaneously on Day 1 of Treatment 1
  Time frame: Treatment 1
- Sitagliptin: Sitagliptin: 100-mg dose of sitagliptin, administered orally, once daily before the LY2189265 dose on Day 1 to Day 5 of Treatment 2.
  Time Frame: Day 1 to Day 5 of Treatment 2
- Sitagliptin + LY2189265: Sitagliptin + LY2189265: 100-mg dose of sitagliptin administered orally, once daily from Day 5 to Day 18 of Treatment 2 in combination with two separate single 1.5-mg doses of LY2189265 administered subcutaneously, immediately prior to the sitagliptin doses on Day 5 and Day 12 of Treatment 2.
  Time Frame: Day 5 to end of Treatment 2
Arm/Group | LY2189265 | Sitagliptin | Sitagliptin + LY2189265
Serious Adverse Events (participants affected / at risk) | 0/26 | 0/29 | 2/29
Other Adverse Events (participants affected / at risk) | 11/26 | 10/29 | 16/29
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | LY2189265 (N=26) | Sitagliptin (N=29) | Sitagliptin + LY2189265 (N=29)
Pneumonia bacterial (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Concussion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Renal failure acute (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | LY2189265 (N=26) | Sitagliptin (N=29) | Sitagliptin + LY2189265 (N=29)
Palpitations (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Chalazion (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Dry eye (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 2 (2)
Dry mouth (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 2 (2) | 0 (0) | 1 (1)
Faeces hard (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Flatulence (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Gingival pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Haematochezia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Lip dry (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (2) | 0 (0) | 4 (6)
Toothache (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 1 (1) | 2 (2)
Fatigue (General disorders) | 3 (3) | 1 (1) | 2 (2)
Feeling jittery (General disorders) | 0 (0) | 0 (0) | 1 (1)
Injection site pain (General disorders) | 2 (2) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 1 (1)
Swelling (General disorders) | 1 (1) | 0 (0) | 0 (0)
Vessel puncture site haematoma (General disorders) | 0 (0) | 1 (1) | 1 (1)
Seasonal allergy (Immune system disorders) | 0 (0) | 1 (1) | 0 (0)
Trichomoniasis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Arthropod bite (Injury, poisoning and procedural complications) | 1 (2) | 0 (0) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 4 (5)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Hypoglycaemia (Metabolism and nutrition disorders) | 1 (2) | 1 (1) | 4 (12)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (2)
Dizziness (Nervous system disorders) | 0 (0) | 1 (4) | 1 (1)
Dizziness postural (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 4 (4) | 1 (1) | 5 (5)
Paraesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Sinus headache (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Somnolence (Nervous system disorders) | 0 (0) | 2 (3) | 0 (0)
Insomnia (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Restlessness (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days